CLINICAL TRIAL: NCT06781034
Title: Descriptive Study on MRI Contrast of Acute Cerebral Hemorrhage in Different Microangiopathies
Acronym: GADO-ICH
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2024/TP-02
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Hemorrhage; Acute Lobar Haematoma
Keywords: Cerebral haemorrhage; MRI
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with acute lobar and deep haematoma: None, pure observational study
  Interventions: Other: None, pure observational study

INTERVENTIONS:
Other: None, pure observational study — None, pure observational study

SUMMARY:
Cerebral haemorrhage represents a minority of acute vascular syndromes (less frequent than ischemic stroke, at around 20%), but with a therapeutic impasse, having no specific treatment.

Arterial contrast ("spot sign") within the hematoma has been described in CT scans as a risk factor for further enlargement and poor prognosis.

An equivalent marker has also been described in gadolinium-enhanced MRI.

By studying the radiological appearance of gadolinium "spot signs" on MRI, which has better parenchymal resolution, the researchers propose to retrace the phenomenology of the acute phase of cerebral hemorrhage in order to better estimate the risk of radiological aggravation by subgroup, which could serve as a target population for future therapeutic trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute cerebral hematomas from existing databases of cerebral amyloid angiopathy and hypertensive microangiopathy managed at Nîmes University Hospital;
* Patients who have undergone a follow-up cerebral CT scan in the event of worsening or for follow-up.

Exclusion Criteria:

* Patient refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute cerebral hematoma from existing databases of cerebral amyloid angiopathy and hypertensive microangiopathy; who underwent a follow-up cerebral CT scan in the event of worsening or for follow-up.
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Presence of spot sign on gadolinium MRI | baseline
  Presence of spot sign on gadolinium MRI (Yes/No)
Morphologic description of gadolinium MRI spot sign | baseline
  morphological (shape, location within the hematoma) description of spot signs on brain MRI
Quantitative description of gadolinium MRI spot sign | baseline
  Quantitative (number and categorial) description of spot signs on brain MRI

SECONDARY OUTCOMES:
association of spot sign with hematoma expansion on follow-up CT | Baseline
  association of spot sign with hematoma expansion on follow-up CT(Yes/No)
Association with the underlaying pathology | Baseline
  Association with the underlaying pathology as identified by the authors (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes

IPD SHARING:
Plan to Share IPD: No